CLINICAL TRIAL: NCT01973296
Title: Implementing an Emergency Department to Home Care Transition Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201200390
Record Dates: First submitted 2013-10-15; First posted 2013-10-31 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: ED Patients With Chronic Medical Illnesses
Keywords: Health Literacy; Care Transition Intervention; Emergency Department Population; Access to Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ED to home care transition (Experimental): The ED to home care transition intervention is a 4-week program that uses a Area Agency on Aging coach to conduct a home visit and three follow up phone calls to help patients develop the skills needed for self-management and to communicate with healthcare providers.
  Interventions: Behavioral: ED to home care transition
- Usual Care (Other): Patients randomized to usual care will receive verbal and written discharge instructions from the treating emergency department physician and nurse as is the standard of care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: ED to home care transition — The CTI coach's role is to build self-management capabilities for the patient and caregiver. During each contact, the coach reviews the four components of the CTI: 1: Follow-up Medical Visit. 2: Knowledge of Red Flag Symptoms. 3: Medication Reconciliation. 4: The Personal Health Record (PHR). The coach assists the patient use the PHR to document and maintain vital information and to communicate with providers.
  Other Names: Care Transition Intervention (CTI)
  Arms: ED to home care transition
Other: Usual Care — Patients randomized to usual care will receive verbal and written discharge instructions from the treating emergency department physician and nurse as is the standard of care.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine whether a new way of educating/coaching chronically ill patients discharged from the Emergency Room will help them receive post-ER health care and strengthen their links to a regular, personal doctor.

DETAILED DESCRIPTION:
Emergency Room (ER) patients with limited health literacy who agree to participate in this study will be asked to complete a survey about how they feel about their health care and how easy or hard it is to get health care. Patients will also be asked for some basic information about themselves like their age, race, gender, employment and marital status, their overall health and health conditions. The research team will review the electronic medical record for information about participants' health conditions and how sick the ER nurse thought the patient was when they came to the ER.

Patients who decide to participate in the study will also be randomly assigned, much like the flip of a coin to receive either a new way of educating patients (the Care Transition Intervention) or normal care. This means:

If patients receive the new way of educating, a coach will visit the patient at home one time one or two days after the ER visit to see how the patient is doing. He/she will talk with the patient about following up with a regular, personal doctor and symptoms to look out for. He/she will help the patient understand their medicines and help the patient make a personal health record. The coach will also tell the patient about the Area Agency on Aging, also called Elder Options. If the patient receives normal care, the patient will not receive a visit from the coach or hear about the Area Agency on Aging but will be given discharge instructions from the ER nurse and doctor.

If the patient receives the new way of educating (the Care Transition Intervention), the coach will call the patient at least 3 times after the ER visit. He/she will talk with the patient about the same items listed above. If the patient receives normal care, the coach will not call. The patient has a 1 in 2 chance of receiving the new way of educating and a 1 in 2 chance of receiving normal care.

All patients will be asked to complete a phone survey 31-60 days after their ER visit. This survey will ask the patient about follow up with a regular, personal doctor. The survey will also ask the patient how they feel about their health care and how easy or hard it is to get health care after an ER visit.

Some patients will also be asked if they are willing to give a separate interview. The study doctor will ask about what happened when you were in the ER. She will also ask about how things went after your ER visit. If the coach contacted you, she will ask about this as well. This interview will be audio recorded.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older,
* are on Medicare,
* are community dwelling,
* reside within the geographical area defined by specific zip codes (to enable home visits),
* have a working telephone, and
* have at least one of the following conditions documented in their medical record: congestive heart failure, chronic obstructive pulmonary disease, coronary artery disease, diabetes, stroke, pneumonia, medical and surgical back conditions (predominantly spinal stenosis), hip fracture, peripheral vascular disease, cardiac arrhythmias, deep venous thrombosis, pulmonary embolism, peptic ulcer disease or hemorrhage.
* health literacy will be assessed with the 66-item Rapid Estimate of Adult Literacy in Medicine (REALM)(Davis, Crouch et al.)

Exclusion Criteria:

* current diagnosis of psychosis,
* active substance abuse related to alcohol or drugs,
* cancer,
* dialysis
* history of organ transplantation,
* have dementia without a live-in caregiver, or
* in hospice care,
* reside outside the defined geographical area,
* reside in a skilled nursing facility, or
* assisted living will be excluded

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Timely and appropriate outpatient medical follow-up | 31-60 days after Emergency Department (ED) visit
  The purpose of this aim is to determine if the ED to home care transition intervention improves patients' access to timely and appropriate outpatient medical follow-up. Patient response to telephone questionnaire will be used to determine time to physician follow-up and type of physician encounter.

SECONDARY OUTCOMES:
Patient activation measure (PAM) level | 31-60 days following ED visit
  The purpose of this aim is to determine if the ED to home care transition intervention improves patients' self management skills as assessed by increased PAM scores.

CONTACTS AND LOCATIONS:
Overall Officials: Donna L Carden, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health, Gainesville, Florida
  - UF Health, Jacksonville, Florida